CLINICAL TRIAL: NCT04454177
Title: SMART TAVR: SMART Watch Facilitated Early Discharge in Patients Undergoing Transcatheter Aortic Valve Replacement
Brief Title: SMART Watch Facilitated Early Discharge in Patients Undergoing Transcatheter Aortic Valve Replacement
Acronym: SMART TAVR
Status: Recruiting | Type: Observational
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-330
Record Dates: First submitted 2020-06-23; First posted 2020-07-01 (Actual); Last update posted 2020-10-27 (Actual); Status verified 2020-06

CONDITIONS: Aortic Stenosis; Valvular Heart Disease; Transcatheter Aortic Valve Replacement
MeSH Terms: conditions — Aortic Valve Stenosis; Heart Valve Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- SMART watch: Medical records from patients aged 18 years or older undergoing Transcatheter Aortic Valve Replacement
  Interventions: Device: HUAWEI watch

INTERVENTIONS:
Device: HUAWEI watch — HUAWEI Watch will be assigned to patients within 24 hours before TAVR. HUAWEI Watch GT series can continuously monitor and record multiple biometric parameters heart rate, step counts, sleep cycles and can detect and record the pulse oxygen saturation, as well as analyze QRS complexes and P waves after triggering.

SUMMARY:
The purpose of this study is to observe conduction disturbance, daily activity level, heart rates, oxygen saturation in patients who underwent Transcatheter Aortic Valve Replacement (TAVR) and to evaluate the utility of the HUAWEI Watch (HUAWEI Technologies Co., Ltd., Shenzhen, China) for the potential early warning sign of changes in multiple biometric parameters including heart rate, rhythm, oxygen saturation, activity, and sleep in patients following TAVR. This will be evaluated in the context of a recently implemented early discharge protocol.

DETAILED DESCRIPTION:
This is a prospective observational cohort study including patients undergoing TAVR procedure in Second Affiliated Hospital of Zhejiang University, School of Medicine. HUAWEI Watch will be assigned to patients within 24 hours before TAVR. HUAWEI Watch GT series can continuously monitor and record multiple biometric parameters heart rate, step counts, sleep cycles and can detect and record the pulse oxygen saturation, as well as analyze QRS complexes and P waves after triggering. The patients will be followed in outpatient clinic visits at 1, 6, 12, 24, and 36 months after TAVR and will commence monitoring with the HUAWEI Watch protocol at least 1 day before the scheduled TAVR procedure to allow familiarity with the device. Patients will be required to activate SMART watch readings (including pulse oxygen saturation and ECG) at least once prior to TAVR and twice per day in the week following TAVR discharge (morning and late afternoon/early evening), at least two days a week for the subsequent month after TAVR discharge and at least once weekly for the remainder of the study. Patients will also be required to activate SMART watch readings at times of any cardiovascular symptoms including dyspnea, chest pain, palpitations, dizziness or presyncope. The health data recorded by HUAWEI Watch will be transmitted to HUAWEI phone application. The Heart Health App (developed by Second Affiliated Hospital, School of Medicine, Zhejiang University) will receive, process and store the data, and transfer it to remote database after approval by patients. A designated heart team member would access the data via a cloud database, contact the patient further investigation or management was deemed necessary.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old;
* Be willing and able to provide informed consent to participate in the study;
* Not share HUAWEI Watch, HUAWEI phone with anyone else;
* Patient has severe aortic stenosis with echocardiographically derived criteria: mean gradient > 40mmHg or maximum velocity greater than 4.0 m/s or an initial aortic valve area of < 1.0 cm2;
* Patient who undergoing elective transfemoral transcatheter aortic valve replacement.

Exclusion Criteria:

* Severe complications of TAVR, such as death, and conversion to SAVR;
* Life expectancy is less than 12 months due to non-heart disease (such as cancer, chronic liver disease, chronic kidney disease, or chronic end-stage lung disease, etc.);
* Severe dementia (cannot sign research informed consent, cannot take care of themselves or complete the study visit);
* The investigator believes that the patient is not suitable to participate in the study or complete the follow-up prescribed by the protocol from other medical, social and psychological aspects;
* The patient is currently participating in another randomized study.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients aged 18 years or older who undergoing Transcatheter Aortic Valve Replacement were the initial target population.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-07-15 (Actual); Primary Completion 2021-08-31 (Estimated); Study Completion 2031-07-01 (Estimated)

PRIMARY OUTCOMES:
Composite of Death and Rehospitalization | 30-day
  Kaplan-Meier Estimate of Death or Rehospitalization from date of discharge, compared to a historical control. Rehospitalization is defined as any hospitalization related to the procedure, the valve or heart failure.
Days Alive and Out of Hospital (DAOH) | 30-day
  Kaplan-Meier Estimate of Days Alive and Out of Hospital (DAOH) from date of discharge, compared to a historical control.

SECONDARY OUTCOMES:
Composite of Death and Rehospitalization | 1-year, 2-year, and 3-year at follow-up
  Kaplan-Meier Estimate of Death or Rehospitalization from date of discharge, compared to a historical control. Rehospitalization is defined as any hospitalization related to the procedure, the valve or heart failure.
Days Alive and Out of Hospital (DAOH) | 1-year, 2-year, and 3-year at follow-up
  Kaplan-Meier Estimate of Days Alive and Out of Hospital (DAOH) from date of discharge, compared to a historical control.
Incidence of pacemaker implantation | 30-day, 6-month, 1-year, 2-year, and 3-year at follow-up
  Incidence of pacemaker implantation.
Time of pacemaker implantation | 30-day, 6-month, 1-year, 2-year, and 3-year at follow-up
  Time of pacemaker implantation will record the time point of the pacemaker implantation.
New York Heart Association (NYHA) Functional Class | baseline, 30-day, 6-month, 1-year, 2-year, and 3-year at follow-up
  NYHA provides a way of classifying the extent of heart failure. New York Heart Association (NYHA) is a functional classification of heart failure based on how much a patient is limited during physical activity. The rating ranges from I-IV, with the NYHA I as no limitation and NYHA IV unable to carry on any physical activity.
Kansas City Cardiomyopathy Questionnaire (KCCQ) | baseline, 30-day, 6-month, 1-year, 2-year, and 3-year at follow-up
  The Kansas City Cardiomyopathy Questionnaire (KCCQ) are on a range of 0-100, in which 100 reflects the best health status and 0 reflects the worst health status.
Hemoglobin | baseline, 30-day, 6-month, 1-year, 2-year, and 3-year at follow-up
  Laboratory examination include hemoglobin, pro-BNP, albumin, creatinine. The unit of Hemoglobin is mg/dL.
Pro-BNP | baseline, 30-day, 6-month, 1-year, 2-year, and 3-year at follow-up
  Laboratory examination include hemoglobin, pro-BNP, albumin, creatinine. The unit of Pro-BNP is pg/mL.
Albumin | baseline, 30-day, 6-month, 1-year, 2-year, and 3-year at follow-up
  Laboratory examination include hemoglobin, pro-BNP, albumin, creatinine. The unit of Albumin is g/L.
Creatinine | baseline, 30-day, 6-month, 1-year, 2-year, and 3-year at follow-up
  Laboratory examination include hemoglobin, pro-BNP, albumin, creatinine. The unit of Creatinine of umol/L.
Echocardiography examinations | baseline, 30-day, 6-month, 1-year, 2-year, and 3-year at follow-up
  Echocardiography examinations include valvular mean gradient, paravalvular leakage, valvular regurgitation, left ventricular ejection fraction, left ventricular diameter, left atrial size, and pulmonary arterial systolic pressure.
Computed tomography examinations | baseline, 30-day, 6-month, 1-year, 2-year, and 3-year at follow-up
  computed tomography examinations include CT assessment parameters, like annular area, perimeter, diameter, SOV, and Coronary height.
Rates of onset of conduction disturbance recorded by Watch | 30-day, 6-month, 1-year, 2-year, and 3-year at follow-up
  Rates of onset of conduction disturbance recorded by Watch
Time of onset of conduction disturbance recorded by Watch | 30-day, 6-month, 1-year, 2-year, and 3-year at follow-up
  Time of onset of conduction disturbance will record the time point of the onset of conduction disturbance.
Rates of onset of new atrial fibrillation or ventricular arrhythmia recorded by Watch | 30-day, 6-month, 1-year, 2-year, and 3-year at follow-up
  Rates of onset of new atrial fibrillation or ventricular arrhythmia recorded by Watch.
Time of onset of new atrial fibrillation or ventricular arrhythmia recorded by Watch | 30-day, 6-month, 1-year, 2-year, and 3-year at follow-up
  Time of new atrial fibrillation or ventricular arrhythmia will record the time point of the onset of new atrial fibrillation or ventricular arrhythmia.
Average daily step counts recorded by Watch | baseline, 30-day, 6-month, 1-year, 2-year, and 3-year at follow-up
  Average daily step counts recorded by Watch is one assessment of daily activity.
Moderate to vigorous physical activity time recorded by Watch | baseline, 30-day, 6-month, 1-year, 2-year, and 3-year at follow-up
  Moderate to vigorous physical activity time recorded by Watch is one assessment of daily activity.
SpO2 detected by Watch | baseline, 30-day, 6-month, 1-year, 2-year, and 3-year at follow-up
  SpO2 detected by Watch
Heart rate assessment recorded by Watch | baseline, 30-day, 6-month, 1-year, 2-year, and 3-year at follow-up
  Heart rate assessment includes average heart rate, resting heart rate, and premature beats ratio recorded by Watch
Assessment of sleep reported by Watch | baseline, 30-day, 6-month, 1-year, 2-year, and 3-year at follow-up
  Assessment of sleep reported by Watch
Rates of cardiac event identified by the watch leading to change of therapy or intervention | 30-day, 6-month, 1-year, 2-year, and 3-year at follow-up
  Rates of cardiac event identified by the watch leading to change of therapy or intervention
Time of cardiac event identified by the watch leading to change of therapy or intervention | 30-day, 6-month, 1-year, 2-year, and 3-year at follow-up
  Time of cardiac event identified by the watch leading to change of therapy or intervention

CONTACTS AND LOCATIONS:
Overall Officials: Jian-an Wang, MD, PhD, Principal Investigator — Second Affiliated Hospital, School of Medicine, Zhejiang University
Locations (1):
- Second Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fan J, Dai H, Guo Y, Xu J, Wang L, Jiang J, Lin X, Li C, Zhou D, Li H, Liu X, Wang J. Smartwatch-Detected Arrhythmias in Patients After Transcatheter Aortic Valve Replacement (TAVR): Analysis of the SMART TAVR Trial. J Med Internet Res. 2024 Jul 19;26:e41843. doi: 10.2196/41843. PMID 39028996
- [Derived] Fan J, Liu Q, Dai H, Zhou D, Guo Y, Xu J, Wang L, Hu P, Jiang J, Lin X, Li C, Liu X, Wang J. Daily Physical Activity Measured by Wearable Smartwatch for Patients Undergoing Transcatheter Aortic Valve Replacement: Insights From the SMART TAVR Study. Circ Cardiovasc Qual Outcomes. 2024 Jan;17(1):e010066. doi: 10.1161/CIRCOUTCOMES.123.010066. Epub 2023 Dec 13. PMID 38088154
- [Derived] Liu X, Fan J, Guo Y, Dai H, Xu J, Wang L, Hu P, Lin X, Li C, Zhou D, Li H, Wang J. Wearable Smartwatch Facilitated Remote Health Management for Patients Undergoing Transcatheter Aortic Valve Replacement. J Am Heart Assoc. 2022 Apr 5;11(7):e023219. doi: 10.1161/JAHA.121.023219. Epub 2022 Mar 29. PMID 35347997